CLINICAL TRIAL: NCT05588258
Title: Comparative, Randomised, Double-blind, Cost-effectiveness Evaluation of Two 10% Urea Creams in Patients With Diabetic Foot Syndrome
Brief Title: Cost-effectiveness Evaluation of Two 10% Urea Creams in Patients With Diabetic Foot Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jose Luis Lazaro Martinez, Prof. Dr., Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21/633-EC_X
Record Dates: First submitted 2022-09-30; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Dosage Forms; Supermarkets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacy cream 10% urea (Active Comparator): Use of pharmacy cream in prevention
  Interventions: Other: Participants were given the 10% urea cream purchased in pharmacy or supermarket as appropriate after randomisation and their foot skin quality was assessed by validated questionnaire.
- Supermarket cream 10% urea (Active Comparator): Use of supermarket cream in prevention
  Interventions: Other: Participants were given the 10% urea cream purchased in pharmacy or supermarket as appropriate after randomisation and their foot skin quality was assessed by validated questionnaire.

INTERVENTIONS:
Other: Participants were given the 10% urea cream purchased in pharmacy or supermarket as appropriate after randomisation and their foot skin quality was assessed by validated questionnaire. — Participants agreed to the interventions after allocation to each arm according to randomisation and after signing an informed consent form. The creams tested in this study provided to participants are authorised for sale within the European Union but are not considered drugs or medical devices. The main purpose of the interventions was based on the care and assessment of the quality of the skin of the participants' feet.
  Other Names: After one month of application of the 10% urea cream assigned after randomisation, the skin quality of the participants' feet was re-evaluated by means of a validated questionnaire.

SUMMARY:
Randomised, double-blind, cost-effectiveness clinical trial of two 10% urea creams purchased in pharmacies and supermarkets in patients with diabetic foot syndrome.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the cost-effectiveness of two 10% urea creams in patients with Diabetic Foot Syndrome.

The methodology was a prospective, longitudinal, single-centre, randomised, double-blind, longitudinal clinical trial that evaluated the skin quality of 20 participating feet belonging to 10 patients with Diabetic Foot Syndrome after the application of two 10% urea creams purchased in pharmacies and supermarkets.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years with Diabetic Foot Syndrome
* Deep or superficial sensory neurological involvement diagnosed by Semmes-Weinstein Monofilament and Rydel-Seiffer tuning fork
* ABI (Ankle Brachial Index) in normal range
* Metabolic Syndrome
* No cognitive impairment
* Patients who agreed to be included in the study by signing a written consent

Exclusion Criteria:

* Patients with hypersensitivity or allergy to any of the components of both creams.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Cost analysis of two 10% urea creams purchased in pharmacies and supermarkets. | 5 months
  The cost analysis will be carried out considering the price per ml of 10% urea cream used by the participants during their participation in the study.
Assessment of the skin quality of participants' feet before and after the cream application intervention using a validated questionnaire. | 5 months
  The assessment of skin quality was carried out using the "Questionnaire for assessment of injury risk and skin quality in patients with diabetic foot syndrome", validated intra-observer and inter-observer by this research group. The minimum score assigned in this questionnaire is 0 points and the maximum score is 12, with higher scores correlating with higher risk of injury and poorer skin quality of the feet.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Lázaro Martínez, Prof. Dr., Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- José Luis Lázaro Martínez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No